CLINICAL TRIAL: NCT06001476
Title: Feasibility and Safety Analysis of Cold Snare Polypectomy in 5-9mm Small Intestinal Polyp Resection in Patients With Peutz-Jeghers Syndrome: A Prospective, Interventional Study
Brief Title: Cold Snare Polypectomy for Small Bowel Polyps in Patients With Peutz-Jeghers Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SDU-QILU-G002
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Peutz-Jeghers Syndrome; Small Bowel Polyp
MeSH Terms: conditions — Peutz-Jeghers Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold snare polypectomy group (Experimental)
  Interventions: Procedure: Cold snare polypectomy

INTERVENTIONS:
Procedure: Cold snare polypectomy — For eligible patients, use cold snare polypectomy to resect 5-9mm short-pedicled, broad-pedicled or sessile small bowel polyps

SUMMARY:
This study aims to evaluate the feasibility and safety of Cold snare polypectomy for removing 5-9mm small intestinal polyps in patients with Peutz-Jeghers Syndrome (PJS),in order to provide some reference for clinical strategy of endoscopic treatment of small intestinal polyps in PJS patients, and may prolong the follow-up period of PJS patients Intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-60, male or female.
* Diagnosed with Peutz-Jeghers Syndrome
* Undergo enteroscopy for small bowel polypectomy.

Exclusion Criteria:

* Absence of at least one study polyp (5-9mm stubby pedicle, wide pedicle and sessile small bowel polyps);
* Be evaluated during enteroscopy for requiring surgical intervention (such as endoscopically difficult to handle giant polyps, intussusception, etc.)；
* With more than 50 polyps ≥1cm found in this enteroscopy examination;
* The polyp has been confirmed to be malignant by pathology, or highly suspicious of malignant transformation under endoscopy;
* Receiving anticoagulant therapy during this treatment;
* Unable or unwilling to provide informed consent.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications in the application of cold snare polypectomy for 5-9mm small bowel polypectomy in patients with PJS | 28 days after the procedure
  The complications include complications during CSP and complications occurring within 28 days after enteroscopy

SECONDARY OUTCOMES:
Incidence of complications during cold snare polypectomy for 5-9mm small bowel polypectomy | Immediately after the procedure
  Including intraoperative bleeding (defined as active haemorrhage for more than 30s), perforation immediately, etc.
Incidence of complications within 28 days after enteroscopy | 28 days after the procedure
  Including Delayed bleeding, delayed perforation, pancreatitis, electrocoagulation syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] van Leerdam ME, Roos VH, van Hooft JE, Dekker E, Jover R, Kaminski MF, Latchford A, Neumann H, Pellise M, Saurin JC, Tanis PJ, Wagner A, Balaguer F, Ricciardiello L. Endoscopic management of polyposis syndromes: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2019 Sep;51(9):877-895. doi: 10.1055/a-0965-0605. Epub 2019 Jul 23. PMID 31342472
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Kawamura T, Takeuchi Y, Asai S, Yokota I, Akamine E, Kato M, Akamatsu T, Tada K, Komeda Y, Iwatate M, Kawakami K, Nishikawa M, Watanabe D, Yamauchi A, Fukata N, Shimatani M, Ooi M, Fujita K, Sano Y, Kashida H, Hirose S, Iwagami H, Uedo N, Teramukai S, Tanaka K. A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study). Gut. 2018 Nov;67(11):1950-1957. doi: 10.1136/gutjnl-2017-314215. Epub 2017 Sep 28. PMID 28970290
- [Background] Sakamoto H, Yamamoto H, Hayashi Y, Yano T, Miyata T, Nishimura N, Shinhata H, Sato H, Sunada K, Sugano K. Nonsurgical management of small-bowel polyps in Peutz-Jeghers syndrome with extensive polypectomy by using double-balloon endoscopy. Gastrointest Endosc. 2011 Aug;74(2):328-33. doi: 10.1016/j.gie.2011.04.001. Epub 2011 Jun 25. PMID 21704992
- [Background] Wang YX, Bian J, Zhu HY, Dong YH, Fang AQ, Li ZS, Du YQ. The role of double-balloon enteroscopy in reducing the maximum size of polyps in patients with Peutz-Jeghers syndrome: 12-year experience. J Dig Dis. 2019 Aug;20(8):415-420. doi: 10.1111/1751-2980.12784. Epub 2019 Jun 17. PMID 31099986
- [Background] Sato J, Hirooka Y, Watanabe O, Nakamura M, Yamamura T, Funasaka K, Ohno E, Kawashima H, Miyahara R, Goto H. Newly Developed Endoscopic Treatment for Small Bowel Polyps: Cold Snare Polypectomy. Intern Med. 2016;55(18):2601-3. doi: 10.2169/internalmedicine.55.6732. Epub 2016 Sep 15. PMID 27629953
- [Background] Hamada K, Takeuchi Y, Ishikawa H, Tonai Y, Matsuura N, Ezoe Y, Ishihara R, Tomita Y, Iishi H. Feasibility of Cold Snare Polypectomy for Multiple Duodenal Adenomas in Patients with Familial Adenomatous Polyposis: A Pilot Study. Dig Dis Sci. 2016 Sep;61(9):2755-9. doi: 10.1007/s10620-016-4165-7. Epub 2016 Apr 28. No abstract available. PMID 27126203
- [Background] Maruoka D, Matsumura T, Kasamatsu S, Ishigami H, Taida T, Okimoto K, Nakagawa T, Katsuno T, Arai M. Cold polypectomy for duodenal adenomas: a prospective clinical trial. Endoscopy. 2017 Aug;49(8):776-783. doi: 10.1055/s-0043-107028. Epub 2017 May 10. PMID 28493238